CLINICAL TRIAL: NCT07214402
Title: Impact of Mediterranean Dietary Intervention on Reactive Oxygen Species Levels and Total Antioxidant Capacity During Pregnancy
Brief Title: Mediterranean Dietary Intervention on ROS Levels and TAC During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Macedonia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 89/19-07-2022
Record Dates: First submitted 2025-09-24; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Healthy Pregnant Women
Keywords: diet; ROS; TAC; oxidative stress; biomarkers; pregnancy; dietary counselling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention on individual dietary counselling about Mediterranean diet (Experimental)
  Interventions: Other: dietary counselling

INTERVENTIONS:
Other: dietary counselling — 12-week antioxidant diet, including increased consumption of antioxidant-rich foods such as ≥5 servings/day vegetables, ≥2 servings/day fruit, ≥8 ½ servings/day wholegrains and 3-4 servings/week lean meat

SUMMARY:
This study focuses on investigating the effects of dietary counseling on antioxidant intakes and how diet can influence reactive oxygen species levels and consequently oxidative stress during pregnancy. This study aims to evaluate oxidative stress biomarkers in pregnant women following online sessions focused on Mediterranean dietary intervention, compared to a control group receiving no dietary guidance. The findings are intended to support the development of targeted public health strategies to reduce the risk of adverse pregnancy outcomes.

DETAILED DESCRIPTION:
At the end of the first trimester of pregnancy (12-13 week of pregnancy), women are randomized into a control group and to intervention group to receive individual dietary counselling. In the intervention group, the dietary counselling about the Mediterranean diet is carried out during 6 online meetings every 15 days and focused on antioxidant nutrients and their intake. They are encouraged to adopt a 12-week antioxidant diet, including increased consumption of antioxidant-rich foods such as ≥5 servings/day vegetables, ≥2 servings/day fruit, ≥8 ½ servings/day wholegrains and 3-4 servings/week lean meat. In the control group, dietary counselling included generic, standard of care guidance about nutrition in pregnancy and is only discussed during a single session. Oxidative stress biomarkers, particularly Reactive Oxygen Species (ROS) and Total Antioxidant Capacity (TAC) levels, are analyzed before and after the study duration in women's serum.

Eight-hour fasting blood samples of all women are collected in evacuated containers with EDTA and without anticoagulant from the cubitus vein, at rest. Samples are centrifuged immediately in a dark room at 500g for 15 min at 4°C. After serum samples are isolated, they are immediately aliquoted and stored at - 80°C until analyzed after specific pretreatments for each assay.

Reactive oxygen species (ROS) are detected in serum using the cell-permeable, ROS-sensitive probe 2',7'-dichlorodihydrofluorescein diacetate (H2DCFDA), which emits fluorescence at 520 nm when oxidized [excitation at 480 nm]. A 0.5 mM stock solution of H2DCFDA in DMSO is used, and the probe is incubated for 30 minutes with human serum samples. ROS levels are assessed at each designated time point. Fluorescence measurements are taken using a Tecan fluorometer with black 96-well microplates. ROS concentrations are quantified in millimolar (mM) units by referencing a standard curve generated using hydrogen peroxide (H2O2) concentrations ranging from 0 to 3 mM.

Trolox equivalent antioxidant capacity methodology is used to evaluate the serum TAC. Antioxidant activity is assayed spectrophotometrically, using a TAC Kit (Total Antioxidant Capacity Colorimetric assay kit, produced by Cayman Chemical Co., Ann Arbor, USA). Antioxidants inhibit the oxidation of 2,2'-azino-bis (3-ethylbenthiazoline)-6-sulphonic acid by the ferryl myoglobin-H2O2 system. Antioxidant concentration is expressed as millimolar Trolox equivalents (mmol/l).

Data are analyzed using IBM SPSS Statistics 19.0. Normality of distribution of data in all groups of pregnant women is determined by Kolmogorov - Smirnov normality test. Descriptive statistics, presented as means ± standard deviations, are performed. An independent samples t-test is conducted to compare the mean baseline levels of ROS between the two groups prior to the intervention, ensuring initial comparability. Baseline non-parametric levels of TAC are compared between the intervention and control groups using the Mann-Whitney U test. The Wilcoxon signed-rank test is used for both variables to compare the two groups after the intervention. Results are considered significant at p < 0.05, with effect sizes (Cohen's d,) reported for clinical relevance.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at the end of the first trimester of pregnancy (12-13 weeks of pregnancy)

Exclusion Criteria:

* Exclusion criteria included hypertension, diabetes, placenta previa, genital tract infections and multiple pregnancies

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Reactive Oxygen Species (ROS) levels will be analyzed before and after the dietary counselling intervention in women's serum and will be quantified in millimolar (mM) units | From enrollment to the end of dietary counselling intervention at 12 weeks
Total antioxidant capacity (TAC) levels will be analyzed before and after the dietary counselling intervention in women's serum and will be expressed as millimolar Trolox equivalents (mmol/l) | From enrollment to the end of dietary counselling intervention at 12 weeks

SECONDARY OUTCOMES:
Weight (in kilograms) berore pregnancy and at the end of the first trimester, as well as height (in meters) will be combined to report BMI (in kg/m^2) berore pregnancy and at the end of the first trimester | From the time before pregnancy to the end of the first trimester of pregnancy (12-13 weeks of pregnancy)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Western Macedonia, Ptolemaida, Greece

IPD SHARING:
Plan to Share IPD: No